CLINICAL TRIAL: NCT05299008
Title: The Effect of Bethanechol on Work of Breathing and Expiratory Tracheal Collapse in Infants With Tracheobronchomalacia Measured by Electrical Activity of the Diaphragm and Bronchoscopy
Brief Title: The Effect of Bethanechol on Tracheobronchomalacia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Charles Preston Pugh, Neonatology Fellow, Arkansas Children's Hospital Research Institute
Other Study IDs: 274192
Record Dates: First submitted 2022-03-18; First posted 2022-03-28 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Tracheobronchomalacia
Keywords: bethanechol; swing Edi; Bronchoscopy
MeSH Terms: conditions — Tracheobronchomalacia | interventions — Bethanechol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants with diagnosis of tracheobronchomalacia treated with bethanechol: Infants with a diagnosis of tracheobronchomalacia by dynamic computed tomography and showing > 50% cross-sectional diameter collapse at 40 to 60 post menstrual age
  Interventions: Drug: Bethanechol

INTERVENTIONS:
Drug: Bethanechol — Infants whom will be treated with bethanechol for tracheobronchomalacia in level IV center Neonatal Intensive Care Unit.
  Other Names: bethanechol chloride

SUMMARY:
The primary aim of this study is to determine if work of breathing estimated using swing Edi will be improved following initiation of bethanechol in infants with tracheobronchomalacia. The investigators hypothesize that work of breathing will be improved in infants with tracheobronchomalacia estimated by a 20% mean decrease in swing Edi following initiation of bethanechol.

DETAILED DESCRIPTION:
Tracheobronchomalacia (TBM) is characterized by dynamic airway collapse resulting from flaccidity of smooth trachealis muscles, and the incidence in infants has been estimated to be as high as 16-50%. Tracheal collapse results in an increase in work of breathing (WOB) which leads to prolonged ventilatory support, increased caloric needs, and prolonged hospitalization. Clinical signs of increased WOB include nasal flaring, increased use of accessory muscles, and paradoxical movements of the rib cage and abdominal wall. Compared with infants with normal airways, infants with TBM have a higher resistive WOB and require increased respiratory support to help attenuate the respiratory work.

Currently, there are no pharmacologic treatment options approved by the Food and Drug Administration for the treatment of TBM. Animal models have shown that muscarinic agonists may improve the tone of the trachealis muscle and airway mechanics. These physiologic improvements have led to the rationale behind use of the long-acting muscarinic agonist, bethanechol, in the treatment of children with tracheomalacia despite no large trials to demonstrate efficacy. By improving trachealis tone and airway mechanics, infants may benefit from an overall decrease in their resistive WOB leading to improved clinical outcomes.

Measurement of actual WOB can be difficult, invasive, and not easily achieved in neonates, however it can be estimated. One method that has been successfully used to estimate WOB in neonates is by swing electrical activity of the diaphragm (Edi) by neurally adjusted ventilatory assist (NAVA). Swing Edi use in NAVA is the difference between the resting tonic activity of the diaphragm (Edi min) and the peak activity of the diaphragm (Edi max) measured by an Edi catheter. By using Swing Edi as a marker for WOB, the investigators propose a methodology to evaluate a physiologic improvement in infants after starting a pharmacologic treatment for TBM.

Though increased WOB is the result of decreased trachealis tone and tracheal collapse, the most accurate method of identifying airway collapse is by direct visualization of the airways. Bronchoscopy is able to give qualitative and semi quantitative impressions of airway collapsibility and has consistently demonstrated a highly favorable safety profile in infants. By performing bronchoscopy before and after bethanechol initiation a direct change may be noted from medical management.

As such, the investigators hypothesize that WOB estimated by swing Edi and tracheal tone identified by direct visualization bronchoscopy will be improved following initiation of bethanechol in infants with tracheobronchomalacia.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a diagnosis of tracheobronchomalacia by dynamic computed tomography and showing > 50% cross-sectional diameter collapse at 40 to 60 post menstrual age and for whom will be treatment with bethanechol in level IV center Neonatal Intensive Care Unit.

Exclusion Criteria:

* Infants with diagnosis of tracheobronchomalacia by dynamic computed tomography with < 50% cross-sectional diameter collapse at 40 to 60 post menstrual age, or infants in which the medical team has not made the decision to start bethanechol.
* Patients with fixed tracheomalacia or bronchomalacia due to external compression of airways.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatient infants in a level IV Neonatal Intensive Care Unit.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary aim of this study is to determine if work of breathing estimated using swing Edi will be improved following initiation of bethanechol in infants with tracheobronchomalacia. | 7 days
  Swing Edi data will be collected continuously by downloading ventilator trends from the 24 hours prior to initiation of bethanechol in infants and subsequently downloaded every 48-72 hours for 7 days after starting bethanechol.

SECONDARY OUTCOMES:
Determining if there is a direct visual change in trachealis tone determined by bronchoscopy following bethanechol initiation in infants with tracheobronchomalacia. | Day 1 and then at 7-14 days
  A baseline flexible bronchoscopy prior to starting of bethanechol followed by a repeat flexible bronchoscopy at days 7-14 of post bethanechol treatment.
Evaluating for change in regional impedance variation by use of Electrical Impedance Tomography | Collect EIT data 24 hours prior to starting bethanechol and on day 7 after starting bethanechol treatment.
  Electrical Impedance Technology (EIT) is a tool used to monitor regional changes in ventilation and lung mechanics.
Evaluating for change in a Pulmonary Severity Score | Data collected 40 weeks to 60 weeks postmenstrual age
  Evaluate a change in a Pulmonary Severity Score (Madden 2005). The pulmonary severity score is defined as the fraction of inspired oxygen (FIO2) x (support) x (medications).
Investigating for change in number of apnea/bradycardia/desaturation events, pain/sedation scores, and doses of sedation medications following bethanechol initiation in infants with tracheobronchomalacia. | Daily from 40 weeks to 60 weeks postmenstrual age
  Data collected 40 weeks to 60 weeks postmenstrual age
Assessing for side effects of bethanechol treatment such an increase in secretions, wheezing, or an increase in loose stools. | 21 days
  Collect the documented effects 7 days before and 14 days after bethanechol initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Charles P Pugh, MD, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenholz SK, Hall RJ, Lilly JR, Shikes RH. Surgical implications of bronchopulmonary dysplasia. J Pediatr Surg. 1987 Dec;22(12):1132-6. doi: 10.1016/s0022-3468(87)80723-6. PMID 3440899
- [Background] Downing GJ, Kilbride HW. Evaluation of airway complications in high-risk preterm infants: application of flexible fiberoptic airway endoscopy. Pediatrics. 1995 Apr;95(4):567-72. PMID 7700760
- [Background] Gunatilaka CC, Higano NS, Hysinger EB, Gandhi DB, Fleck RJ, Hahn AD, Fain SB, Woods JC, Bates AJ. Increased Work of Breathing due to Tracheomalacia in Neonates. Ann Am Thorac Soc. 2020 Oct;17(10):1247-1256. doi: 10.1513/AnnalsATS.202002-162OC. PMID 32579852
- [Background] Wagner EM, Jacoby DB. Methacholine causes reflex bronchoconstriction. J Appl Physiol (1985). 1999 Jan;86(1):294-7. doi: 10.1152/jappl.1999.86.1.294. PMID 9887142
- [Background] Bass R, Santiago M, Smith L, Quinlan C, Panitch H, Giordano T, Piccione J. (2018). Bethanechol in Tracheomalacia: Two Case Series and a Review of the Literature. Pediatric Allergy, Immunology, and Pulmonology. 31:3, 180-183. https://doi.org/10.1089/ped.2018.0880
- [Background] Bhutani VK, Koslo RJ, Shaffer TH. The effect of tracheal smooth muscle tone on neonatal airway collapsibility. Pediatr Res. 1986 Jun;20(6):492-5. doi: 10.1203/00006450-198606000-00002. PMID 2872649
- [Background] Panitch HB, Keklikian EN, Motley RA, Wolfson MR, Schidlow DV. Effect of altering smooth muscle tone on maximal expiratory flows in patients with tracheomalacia. Pediatr Pulmonol. 1990;9(3):170-6. doi: 10.1002/ppul.1950090309. PMID 1980538
- [Background] Hysinger E, Friedman N, Jensen E, Zhang H, Piccione J. Bronchoscopy in neonates with severe bronchopulmonary dysplasia in the NICU. J Perinatol. 2019 Feb;39(2):263-268. doi: 10.1038/s41372-018-0280-y. Epub 2018 Dec 5. PMID 30518799
- [Background] Madan A, Brozanski BS, Cole CH, Oden NL, Cohen G, Phelps DL. A pulmonary score for assessing the severity of neonatal chronic lung disease. Pediatrics. 2005 Apr;115(4):e450-7. doi: 10.1542/peds.2004-1293. PMID 15805348
- [Background] Nealon E, Rivera BK, Cua CL, Ball MK, Stiver C, Boe BA, Slaughter JL, Chisolm J, Smith CV, Cooper JN, Armstrong AK, Berman DP, Backes CH. Follow-up after Percutaneous Patent Ductus Arteriosus Occlusion in Lower Weight Infants. J Pediatr. 2019 Sep;212:144-150.e3. doi: 10.1016/j.jpeds.2019.05.070. Epub 2019 Jun 28. PMID 31262530
- [Background] Lee J, Kim HS, Jung YH, Shin SH, Choi CW, Kim EK, Kim BI, Choi JH. Non-invasive neurally adjusted ventilatory assist in preterm infants: a randomised phase II crossover trial. Arch Dis Child Fetal Neonatal Ed. 2015 Nov;100(6):F507-13. doi: 10.1136/archdischild-2014-308057. Epub 2015 Jul 15. PMID 26178463
- [Background] Bergeron M, Cohen AP, Cotton RT. The Management of Cyanotic Spells in Children with Oesophageal Atresia. Front Pediatr. 2017 May 15;5:106. doi: 10.3389/fped.2017.00106. eCollection 2017. PMID 28555179
- [Background] Masters IB, Zimmerman PV, Pandeya N, Petsky HL, Wilson SB, Chang AB. Quantified tracheobronchomalacia disorders and their clinical profiles in children. Chest. 2008 Feb;133(2):461-7. doi: 10.1378/chest.07-2283. Epub 2007 Nov 7. PMID 17989148
- [Background] Wallis C, Alexopoulou E, Anton-Pacheco JL, Bhatt JM, Bush A, Chang AB, Charatsi AM, Coleman C, Depiazzi J, Douros K, Eber E, Everard M, Kantar A, Masters IB, Midulla F, Nenna R, Roebuck D, Snijders D, Priftis K. ERS statement on tracheomalacia and bronchomalacia in children. Eur Respir J. 2019 Sep 28;54(3):1900382. doi: 10.1183/13993003.00382-2019. Print 2019 Sep. PMID 31320455
- [Background] DeBoer EM, Prager JD, Kerby GS, Stillwell PC. Measuring Pediatric Bronchoscopy Outcomes Using an Electronic Medical Record. Ann Am Thorac Soc. 2016 May;13(5):678-83. doi: 10.1513/AnnalsATS.201509-576OC. PMID 26816220
- [Background] Su YT, Chiu CC, Lai SH, Hsia SH, Lin JJ, Chan OW, Chiu CY, Tseng PL, Lee EP. Risk Factors for Tracheobronchomalacia in Preterm Infants With Bronchopulmonary Dysplasia. Front Pediatr. 2021 Jun 25;9:697470. doi: 10.3389/fped.2021.697470. eCollection 2021. PMID 34249821